CLINICAL TRIAL: NCT06861296
Title: Effect of Postpartum Hemorrhage Education Structured With Flipped Learning Model on Knowledge, Skills, Clinical Self-Efficacy and Satisfaction of Midwifery Students
Brief Title: Flipped Learning in PPH Education: Impact on Midwifery Students' Knowledge, Skills, Self-Efficacy, and Satisfaction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Sumeyra Damsarsan, Lecturer, Saglik Bilimleri Universitesi
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 913715751 2025/09
Record Dates: First submitted 2025-01-28; First posted 2025-03-06 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Teaching Innovation; Midwifery Students Education; Postpartum Hemorrhage; Flipped Classroom Model in Teaching
Keywords: Flipped Learning; Postpartum Hemorrhage; Midwifery Education; Clinical Self-Efficacy
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Masking Description: The person who assessed the students' knowledge and skills and the person who performed the statistical analysis were blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Traditional Education Model Based Education Group) (No Intervention): This group will be trained with the traditional education model regarding the management of postpartum hemorrhage. Theoretical training in this group is planned as face to face in the classroom with the traditional lecture model; practical training is planned as face to face in the laboratory.
- Intervention Group (Flipped Learning Model Based Training Group) (Experimental): This group will receive training on postpartum hemorrhage management using the reverse learning model. Theoretical and practical lessons will be given primarily through out-of-class activities. Students will learn simple basic information outside of class whenever they want with the instructor's videos. Thus, advanced methods (gamification, concept analysis, group discussions) can be applied to ensure active and permanent learning in in-class activities.
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — (Flipped Learning Model Based Training Group)-Arm Description: This group will receive training on postpartum hemorrhage management using the reverse learning
  Arms: Intervention Group (Flipped Learning Model Based Training Group)

SUMMARY:
Maternal death refers to a woman's death due to direct or indirect causes during pregnancy, childbirth, or within 42 days postpartum. Postpartum hemorrhage (PPH) is the leading cause of maternal mortality globally and in our country. Rapid and effective management of PPH is crucial in reducing maternal deaths. WHO, UNFPA, and UNICEF emphasize the critical role of midwives in PPH management, highlighting the importance of enhancing their knowledge and skills during pre-graduate education.

Traditional education models are often insufficient for fostering permanent learning, especially in acquiring psychomotor skills like PPH management. In traditional learning, classroom instruction follows a teacher-centered approach, covering only the first two levels of Bloom's taxonomy-knowledge and comprehension-while higher-order cognitive skills such as application, analysis, synthesis, and evaluation are left to individual effort. However, effective and lasting learning requires an active learning environment where students engage more deeply with the material.

The flipped learning model addresses these challenges by allowing students to access foundational knowledge outside the classroom and dedicate class time to higher-order skills like discussion, application, and problem-solving. This model enhances learning through technology and interactive face-to-face activities, fostering professional competence in health education. While the flipped learning model is widely used in health education, most studies focus on theoretical knowledge, with limited research on psychomotor skill acquisition.

To our knowledge, this study is the first to evaluate the effectiveness of flipped learning in midwifery education for both theoretical and psychomotor skill development. The findings are expected to contribute to advancements in midwifery education and healthcare services.

ELIGIBILITY:
Inclusion Criteria:

* Being a 3rd year student in the Midwifery Department of Gülhane Health Sciences Faculty
* Having successfully completed the normal birth course
* Agreeing to participate in the study

Exclusion Criteria:

* Students who were on sick leave or on sick leave during the study period
* Those who did not take the normal birth course or failed
* Students who were absent from at least one session of the training program

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum Hemorrhage Knowledge and Skills | Baseline (just before training) and 3 weeks after the completion of training.
  Description: Knowledge and skills related to postpartum hemorrhage will be assessed.
  Assessment Tool: A test developed by researchers, with scoring determined based on expert opinions.
  Unit of Measure: Test score (numerical). (Scoring for this test will be determined after the tests are developed by the researcher and expert opinions are received.)
Clinical Skills Self-Efficacy | At the beginning (immediately before the practical training) and 3 weeks after the completion of the practical training.
  Description: The self-efficacy levels of students regarding clinical skills will be evaluated.
  Assessment Tool: Clinical Skills Self-Efficacy Scale. The minimum score is 14, and the maximum score is 70. Higher scores indicate greater self-efficacy.
  Unit of Measure: Scale score (range: 14-70).
Educational Satisfaction | After the theoretical and practical training has been fully completed for both groups (approximately 10-14 weeks after the start of the training)
  Description: Students' satisfaction with postpartum hemorrhage training will be measured, comparing traditional education with the flipped learning model.
  Assessment Tool: A satisfaction scale rang. The minimum score is 10 and the maximum score is 0. Higher scores indicate greater educational satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The results of this study will be published in the form of a thesis, articles, and conference presentations. De-identified individual participant data (IPD) may be shared upon request, in accordance with appropriate ethical principles.
Supporting Information: CSR
Time Frame: After completion of the study (approximately 1 year later)
Access Criteria: Researchers who wish to access the data should submit a formal request, providing details of their research purpose. Data sharing will be considered in compliance with ethical guidelines and institutional policies.